CLINICAL TRIAL: NCT02265861
Title: The Higher Response of Vascular Endothelial Growth Factor and Angiotensin-II to Human Chorionic Gonadotropin in Women With Polycystic Ovary Syndrome
Brief Title: Response of VEGF and AT-II to HCG in PCOS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Wang Yong, Associate Professor, Nanjing University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: NanjingUSMwy
Record Dates: First submitted 2014-10-03; First posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome; Vascular endothelial growth factor; Angiotensin-Ⅱ; Ovarian hyperstimulation syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome; Ovarian Hyperstimulation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): typical PCOS
  Interventions: Drug: HCG
- Group 2 (Experimental): PCOS without PCO
  Interventions: Drug: HCG
- Group 3 (Experimental): PCOS without HA
  Interventions: Drug: HCG
- Group 4 (Experimental): Control
  Interventions: Drug: HCG

INTERVENTIONS:
Drug: HCG

SUMMARY:
This research is to investigate the response of vascular active factors, vascular endothelial growth factor (VEGF) and angiotensin-Ⅱ (AT-Ⅱ) to ovary stimulation during 24h in patients with polycystic ovary syndrome (PCOS).Controled prospective clinical study involved 60 women undergoing in vitro fertilization. Fifty-two patients with PCOS and 8 control cases were stimulated with human chorionic gonadotropin (HCG) during the early follicular phase of the menstrual cycle (4st to 7th days of the cycle).The blood was sampled before the injection (0 hour) and at the 3, 6, 12, 18 and 24 hours points after the stimulation. VEGF, AT-Ⅱ were measured by radioimmunoassay.

DETAILED DESCRIPTION:
After ovary stimulation, the level of VEGF in typical PCOS patients is obviously increased at the 3hs time point (p<0.05), while there is no difference with VEGF at all other time point among the four groups. As for AT-Ⅱ, before and after the ovary stimulation, at all time points, the AT-Ⅱ levels in serum of patients with different phenotypes of PCOS by Rotterdam criteria are all higher than the controls without PCOS. After the ovary stimulation, AT-Ⅱ in typical PCOS patients is obviously increased at 3hs time point, p<0.05. The response of VEGF and AT-Ⅱ to HCG in women with typical PCOS is higher in 24 hours after the stimulation during the early follicular phase. The response to the stimulation is different in patients with different phenotypes of PCOS by Rotterdam criteria. Serum VEGF and AT-Ⅱ levels as a possible contributor to a great risk of developing OHSS in patients with typical PCOS during the early follicular phase in 24 hours after the ovary stimulation.

ELIGIBILITY:
Inclusion Criteria:

* A total of 60 women were recruited and divided into four groups by Rotterdam criteria according to three typical characters:

  1. biochemical characteristics of hyperandrogenism (HA)
  2. chronic anovulation
  3. polycystic ovary morphology (PCO).

Exclusion Criteria:

* All women were matched for age (<35 yr).
* All subjects were screened, and no other endocrine disturbances (thyroid, adrenal) or medical illnesses were found.
* All the patients did not have any hormonal preparation during the 3 months preceding the study.

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Levels of vascular endothelial growth factor(VEGF) and angiotensin-Ⅱ(AT-Ⅱ) | 24 hours

REFERENCES:
- [Derived] Qu J, Che Y, Xu P, Xia Y, Wu X, Wang Y. The Higher Response of Vascular Endothelial Growth Factor and Angiotensin-II to Human Chorionic Gonadotropin in Women with Polycystic Ovary Syndrome. Int J Fertil Steril. 2015 Jan-Mar;8(4):373-8. doi: 10.22074/ijfs.2015.4176. Epub 2015 Feb 7. PMID 25780518